CLINICAL TRIAL: NCT01895725
Title: Correlation of Artherosclerotic Plaque Volume and Intima Media Thickness With Soluble P-selectin
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Peter Marschang, Prof. MD, Medical University Innsbruck
Other Study IDs: P-selectin 03-13
Record Dates: First submitted 2013-06-28; First posted 2013-07-10 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Cardiovascular Risk Factors; Coronary Artery Disease; Cerebrovascular Disease; Peripheral Artery Disease
MeSH Terms: conditions — Coronary Artery Disease; Cerebrovascular Disorders; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The proposed project is a prospective observational, single-center cohort study aimed to examine the progression of atherosclerotic alterations of the carotid arteries (IMT, plaque volume) during a follow-up of up to four years and to correlate the observed changes with traditional and novel biomarkers of atherosclerosis. A total of 600 subsequent patients with or established cardiovascular disease or at least one cardiovascular risk will be tested with a high-frequency ultrasound probe equipped with automated IMT measurements and 3D quantitative plaque volumetry. Plasma samples will be collected and tested for traditional and novel cardiovascular risk factors. Both ultrasound examinations and blood sampling will be repeated once per year to assess changes in these parameters over time depending on treatment modalities, which are left to the discretion of the treating physicians. The primary endpoint of the planned study will be the correlation between P-selectin and the progression of atherosclerosis as measured by plaque volume and IMT in the carotid and femoral arteries, respectively. Secondary endpoints will include the correlation of established (hypertension, smoking, diabetes, dyslipidemia) and novel risk factors (hsCRP, P-selectin, cholesteryl ester transfer protein (CETP), intercellular adhesion molecule-1 (ICAM-1), CETP TaqIb polymorphism) with the progression of atherosclerosis, the correlation of cardiovascular events with the progression of atherosclerosis and the additional predictive value of plaque volume and IMT compared to an established risk score (SCORE card).

ELIGIBILITY:
Inclusion Criteria:

* Patients (male and female) aged 30 to 85 years
* with at least one traditional cardiovascular risk factor (hypertension, smoking, diabetes, dyslipidemia, family history) or established coronary artery disease, cerebrovascular disease, or peripheral artery disease diagnosed by objective testing

Exclusion Criteria:

* lack of informed consent
* the impossibility of follow-up testing once per year for the following four years

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to ultrasound examinations of the carotid and/or femoral arteries for standard indications will be screened for potential inclusion into the study
Sampling Method: Non-Probability Sample
Enrollment: 443 (Actual)
Dates: Start 2013-06; Primary Completion 2020-01-30 (Actual); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between P-selectin and the progression of atherosclerosis | up to 4 years
  The primary endpoint of the planned study will be the correlation between P-selectin and the progression of atherosclerosis as measured by plaque volume and IMT in the carotid and femoral arteries

SECONDARY OUTCOMES:
Correlation of cardiovascular events with the progression of atherosclerosis | up to 4 years
  As secondary endpoints, cardiovascular events (cardiovascular death, myocardial infarction, percutaneous transluminal coronary angioplasty (PTCA), coronary bypass surgery, stroke, transient ischemic attack (TIA), surgery for aortic aneurysm, critical limb ischemia, peripheral percutaneous transluminal angioplasty (PTA), peripheral bypass) will be correlated with the progression of atherosclerosis and the additional predictive value of plaque volume and IMT in carotid and or femoral arteries compared to an established clinical risk score risk score (SCORE card) will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Peter Marschang, MD, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Department for Internal Medicine III, Innsbruck, Austria